CLINICAL TRIAL: NCT04095091
Title: Real-time Tumor Localization and Guidance for Radiotherapy Using Ultrasound (US) and Magnetic Resonance (MR)
Status: Terminated | Type: Observational
Why Stopped: Device to be used in study is no longer available
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-0684; R01CA190298-01A1 (NIH); A534800 (Other: UW Madison); SMPH\MEDICAL PHYSICS (Other: UW Madison); Protocol Version 5/27/2021 (Other: UW Madison)
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Tumor, Solid
Keywords: Radiotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control Group: Healthy volunteers will be asked to complete a single imaging session that will include acquiring simultaneous 4D ultrasound and 4D MRI scan.
  A substudy including patients undergoing radiotherapy for malignancies of the abdomen and pelvis. They will also be asked to complete a single imaging session that will include acquiring simultaneous 4D ultrasound and 4D MRI scan.
  Interventions: Device: 4D Planar US Transducer
- Patient Group: Patients receiving radiotherapy for malignancies of the abdomen and pelvis will be asked to complete two research visits lasting approximately one hour. Each visit will include a 30 minute combined 4D ultrasound and 4D MRI scan.
  Interventions: Device: 4D Planar US Transducer

INTERVENTIONS:
Device: 4D Planar US Transducer — This 4D planar US transducer is being developed and validated to provide a novel image-guidance technique to directly track tumor motion during radiation therapy that is coupled to a pre-treatment calibration training image set consisting of a simultaneous 4D ultrasound and 4D magnetic resonance imaging (MRI) acquisition.
  Other Names: 4D US

SUMMARY:
The primary objective of this protocol is to evaluate the feasibility of acquiring simultaneous 4D ultrasound and 4D MRI scans. The imaging performance of the US and MRI scans will be characterized. The secondary objective of this study is to determine if several salient features identified in the US scan can be used to predict target motion identified in the MR scan.

DETAILED DESCRIPTION:
The goal of radiotherapy treatment of cancer is to cure or locally control the disease while minimizing complications to healthy tissue. Given the complexity of tumor and normal tissue response to radiation, precise and accurate delivery of absorbed dose distributions, within known tolerances, is necessary to achieve the maximum therapeutic ratio. The complex treatment process of radiotherapy introduces geometrical uncertainties including respiratory induced tumor motion. The goal of this research is to develop and validate a novel image-guidance technique to directly track tumor motion using a 4-dimensional (4D) planar ultrasound (US) transducer during radiation therapy that is coupled to a pre-treatment calibration training image set consisting of a simultaneous 4D ultrasound and 4D magnetic resonance imaging (MRI) acquisition. The image sets will be rapidly matched using advanced image and signal processing algorithms, allowing the display of virtual MR images of the tumor/organ motion in real-time from an ultrasound acquisition.

ELIGIBILITY:
Inclusion Criteria (Healthy Volunteers):

* Must be eighteen (18) years of age or older.
* Must be able to provide informed consent.

Inclusion Criteria (Patients):

* Patients diagnosed with malignancies of the liver.

Exclusion Criteria (All):

* Under the age of eighteen (18) years.
* BMI exceeds the size of the bore of the MRI scanner.
* Unable or unwilling to provide informed consent.
* Contraindications, as described in the volunteer consent form, to MR or US scanning such as but not limited to accidental or implanted ferrous metal and/or implanted devices whose function can be disturbed by the main magnetic field, gradient magnetic fields, or radiofrequency energy.
* Women who are pregnant, suspect they might be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be recruited from the general population. Patients will be recruited from clinics that serve this patient population.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Feasibility testing | 12 Months
  To conduct non-contrast agent MR and ultrasound scans in order to evaluate and demonstrate, on a continuing basis, the technical and clinical feasibility of new or modified features (the "Prototype") of a combined MRI and ultrasound system, and software. Prototype MRI and ultrasound systems are defined as components of the MRI system (software) and ultrasound system (hardware and software) that have been modified in some form.
MR/US Motion Management Platform | 12 Months
  The goal of this trial is to assess the feasibility of implementing the system into clinical practice and to compare the dosimetric advantages of its use. In a retrospective analysis, the patients' standard treatment plan with international target volume (ITV) expansion will be directly compared with a second treatment plan using a smaller respiratory-gated margin (i.e., gross tumor volume (GTV)-only expanded for planning target volume (PTV) without ITV expansion). Normal tissue constraints will be specified and follow standard clinical constraints. The percent of liver volume receiving greater than 18 Gy will be used as a quantitative metric to assess the dosimetric impact of our platform. In addition, overall treatment time with the relative "beam on time" and duty cycle will also be compared. Additionally, the ultrasound acquisition during treatment will be used to assess intra- and interfraction changes in breathing patterns as the patients progress through treatment.

SECONDARY OUTCOMES:
Accuracy of image-guidance technique | 12 Months
  The accuracy of our image-guidance technique will be done by showing that several salient features identified in the US scan can be used to predict/model target motion identified in the MR scan. In this context the target will be a large easily identifiable structure in the test subject (e.g. cyst, vessel). MRI and ultrasound images will be acquired simultaneously such that the motion of tissues or organs in the body can be effectively tracked as a function of respiratory state in the subject. In this manner, the ultrasound system will allow real-time tracking of salient features in the patient that are indicative of the respiratory state.
Test/re-test | 12 Months
  A secondary objective of this substudy is to evaluate the accuracy of probe re-position during subsequent treatment sessions (i.e. test/re-test) in cancer patient subjects. The probe will be positioned during one of the patient subjects and images will be acquired. During a subsequent treatment session the probe will be re-positioned and images will be acquired. The image data will be used to evaluate to measure the concordance between the two datasets.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Bednarz, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States